CLINICAL TRIAL: NCT01025895
Title: Anterior Cruciate Ligament (ACL) Reconstruction: Single Bundle Versus Double Bundle
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 144/09
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-07

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: arthroscopic surgical procedure
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

ARMS (2):
- single bundle (Active Comparator): acl reconstruction - single bundle technique
  Interventions: Procedure: acle reconstruction - single bundle technique
- double bundle (Experimental): acl reconstruction - double bundle technique
  Interventions: Procedure: acl reconstruction - double bundle technique

INTERVENTIONS:
Procedure: acl reconstruction - double bundle technique
  Arms: double bundle
Procedure: acle reconstruction - single bundle technique
  Arms: single bundle

SUMMARY:
ACL tear is a common injury among athletes. The recommended treatment includes reconstruction of the ligament. The common reconstruction technique is single bundle reconstruction. However, this technique does not simulate the natural structure of the ligament. The purpose of the study is to compare between the common procedure, Single Bundle reconstruction with the Double Bundle reconstruction technique.

ELIGIBILITY:
Inclusion Criteria:

* knee instability with a history of ACL tear
* diagnosed ACL tear according to MRI
* age range 16-40.

Exclusion Criteria:

* previous surgery in the knees
* multiple ligament raptures
* partial ACL tear
* severe cartilage degeneration
* genovaruse/genovalgus
* thin hamstrings tendons
* oper epiphysis in the knee joint
* patient with muscle/neurological problem that increases the tendency to fall

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
WOMAC, VAS, SF-36, Lisholm, Knee society score, isokinetic muscle strength testing, Single HOP test , Tripple Hop Test | pre-op. 1 day post op., 7-14 days post op., 6 weeks post op., 12 weeks post op., 26 weeks post op., 1 year post op., 2 years post op.